CLINICAL TRIAL: NCT04197245
Title: Efficacy of Saline Injection Therapy in Atrophic Acne Scars: A Clinical Trial in a Tertiary Care Hospital of Karachi
Brief Title: Efficacy of Saline Injection Therapy in Atrophic Acne Scars
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Sidra Khan, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2018-GENL/9008/JPMC
Record Dates: First submitted 2019-12-06; First posted 2019-12-13 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Atrophic; Scars
Keywords: Acne; Scars; DLQI
MeSH Terms: conditions — Atrophy; Cicatrix; Acne Vulgaris | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- group on treatment (Experimental): saline injection has been given intradermal in atrophic scars of acne on face.
  Interventions: Drug: saline injection therapy in post-acne atrophic scars

INTERVENTIONS:
Drug: saline injection therapy in post-acne atrophic scars — saline injection contains 0.9% isotonic sodium chloride solution
  Other Names: normal saline, isotonic saline

SUMMARY:
The purpose of the study was to determine the efficacy of saline injection in post-acne atrophic scars on face. All patients with mild, moderate & severe post-acne atrophic scars, above age of 15 years without any co-morbid conditions were included in the study. After giving local anesthesia, the isotonic saline solution has been administered intra- and sub-dermally in post-acne atrophic scars on face. The sessions were done weekly, for 12 weeks. The results were assessed by the photographs, sharquie scoring system & Dermatology Life Quality Index score at the start and at the end of the treatment. SPSS 23 was used to analyze the data. The analysis of data showed that the response of saline injection was significant in mild and moderate scars, without any significant side effects.

DETAILED DESCRIPTION:
The study was conducted for the determination of saline injection effectiveness in post-acne atrophic scars in patients referred to the department of dermatology in Jinnah postgraduate medical centre, Karachi, Pakistan from January 2019 to July 2019, after receiving approval letter from the institutional ethical and research committee of the hospital.

Forty-nine patients were selected after calculating the sample size through the NCSS software. The patients were selected with the age ranging from 15-35years of either gender, after excluding hypertension, cardiovascular disorders, pregnancy, lactation & hypersensitivity to lidocaine. The procedure has been explained to each patient & written consent was taken. Before starting treatment, the photographs were taken for each patient with their permission & sharquie scoring system for grading scars and Dermatology Life Quality Index scores were calculated.

During each session, after all sterilization techniques, patient has been pain-free with the application of local anesthesia, then 0.9% isotonic saline is injected intra- and sub-dermally in post-acne atrophic scars with 1cc syringe of 30-gauge needles, on both sides of face. The volume of saline injected depends upon the numbers, width and depth of the individual scars. It has been injected up to scar elevation by overfilling with saline & spreading into surrounding tissue as well.

A total of 12 sessions were done weekly. The efficacy of treatment has been assessed by comparing photographs, sharquie scoring system for grading scars and Dermatology Life Quality Index scores at the start and at the end of treatment.

The sharquie scoring system for grading scars has been calculated through assessing number of scars, proportion of the area of the face involved, morphology of scars including color or type and social behavior of the patient. The final scores obtained by adding all scores, were compared with the initial ones, at the end of treatment.

The Dermatology Life Quality Index (DLQI) has been calculated through simple questionnaire, consisting of 10 questions related to the effect of disease and its treatment on the daily activities of patient and the impact on the social behavior of the patient towards friends and relatives. DLQI scores has been interpreted, regarding the effect on patients' life as follows:

* 0-1 = No effect
* 2-5 = Small effect
* 6-10 = Moderate effect
* 11-20 = Very large effect
* 21-30 = Extremely large effect

At the end of treatment, results were compared to assess the improvement in everyday activities and social behaviors of the patients.

The evaluation of result was done by SPSS version 23. The side effects were also assessed regarding erythema, itching , pain & dys-pigmentation.

In this study three patients of post-acne atrophic scars also had atrophic scars due to trauma in the childhood, on their face. On the request of the patients, these scars were also filled with saline injection, in addition to their post-acne atrophic scars.

During treatment, change in the post-acne pigmentation, skin tightening, eruption of new acne lesions, healing of old lesions has also been observed.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 15years
* Maximum age 35 years
* Both males and females with mild, moderate and severe post-acne atrophic scars on face.

Exclusion Criteria:

* Hypertension
* Cardiovascular disorders
* Pregnancy
* Lactation
* Hypersensitivity to lidocaine.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
change in morphology of scars | 12 weeks
  there is significant change in the morphology of scars, assessed by sharquie score for grading scars

SECONDARY OUTCOMES:
change in dermatology life quality index of patients | 12 weeks
  significant change in dermatology life quality index of patients

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ghafoor, FCPS, Study Director — jinnah postgraduate medical centre, karachi
Locations (1):
- Jinnah postgraduate medical centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Dhalimi M, Jaber A. Treatment of atrophic facial acne scars with fractional Er:Yag laser. J Cosmet Laser Ther. 2015;17(4):184-8. doi: 10.3109/14764172.2015.1007067. Epub 2015 Feb 13. PMID 25588037
- [Result] Bagherani, N, Smoller, B. Introduction of a novel therapeutic option for atrophic acne scars: saline injection therapy. Global dermatology. 2015;2(6): 225-7
- [Result] Hazarika N, Archana M. The Psychosocial Impact of Acne Vulgaris. Indian J Dermatol. 2016 Sep-Oct;61(5):515-20. doi: 10.4103/0019-5154.190102. PMID 27688440